CLINICAL TRIAL: NCT02345187
Title: Impact of a Multiple Micronutrient (MMN) Fortified Powder Supplemented With Bacopa Monnieri Extract (EBM) on Hemodynamic Responses as Measured by Functional Magnetic Resonance Imaging (fMRI) in Indian School Children (11-12 Yrs; Inclusive) After Approximately 4 Months of Intervention: an Exploratory, Randomized, Double-blind, Controlled Trial
Brief Title: fMRI Study to Investigate Hemodynamic Changes in Brain Resulting From Supplementation of Bacopa Monnieri Extract and Multiple Micronutrient Supplementation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Mahajan Imaging Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 202191; RH02384 (Other: GSK)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Growth and Development

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Active Comparator): Entire content of a sachet of the beverage powder fortified with multiple micronutrients and bacopa monnieri extract will be emptied in a graduated drinking tumbler and reconstituted with 180 mL potable lukewarm water. Water will be added to the tumbler gradually with stirring to avoid lump formation. The reconstituted beverage will be administered to the participants orally twice daily for 17 weeks
  Interventions: Dietary Supplement: Beverage powder fortified with Bacopa Monnieri Extract and Multiple Micronutrient supplementation
- Control arm (Placebo Comparator): Entire content of a sachet of the non-fortified isocaloric beverage powder will be emptied in a graduated drinking tumbler and reconstituted with 180 mL potable lukewarm water. Water will be added to the tumbler gradually with stirring to avoid lump formation. The reconstituted beverage will be administered to the participants orally twice daily for 17 weeks
  Interventions: Dietary Supplement: Non-fortified isocaloric beverage powder

INTERVENTIONS:
Dietary Supplement: Beverage powder fortified with Bacopa Monnieri Extract and Multiple Micronutrient supplementation — The study product (fortified beverage powder reconstituted with 180 mL lukewarm water) will be administered twice daily for 17 weeks
  Arms: Treatment Arm
Dietary Supplement: Non-fortified isocaloric beverage powder — The study product (non-fortified isocaloric beverage powder reconstituted with 180 mL lukewarm water) will be administered twice daily for 17 weeks
  Arms: Control arm

SUMMARY:
The study will aim to compare the effects of a beverage powder fortified with multiple micronutrients and Bacopa monnieri extract (test product) to a non-fortified isocaloric beverage powder (control product) on cognitive outcomes of attention and working memory.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent from participant's parents/ legally acceptable representative (LAR) and voluntary written assent from the subject and a signed, dated copy of the informed consent and assent forms.
* Right handed, School going children (participants) aged 11-12 years, inclusive
* Satisfactory completion of baseline imaging scan basis participant's ability to stay still, with acceptable MRI/fMRI image quality as determined by technical expert at the imaging centre
* Compliance of participant and participant's parents/LAR with all study procedures and restrictions.
* Participant is able to read and comprehend one of the languages used for cognitive assessment (English or Hindi)
* Participant with Z-scores of Body Mass Index (BMI) for age of >-2 to <+1

Exclusion Criteria:

* Child in Care (CiC); A child who has been placed under the control or protection of an agency, organization, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. A CiC does not include a child who is adopted or has an appointed legal guardian.
* Known or suspected intolerance or hypersensitivity to the study materials, any of their stated ingredients or any known food allergies like nut allergy, gluten allergy or lactose intolerance.
* Severe anemia with hemoglobin<8g/Dl, Attention Deficit Hyperactivity Disorder (ADHD), reading dyslexia or any other behavioral disorder.
* Participation in another clinical study or receipt of an investigational drug within 30 days prior to the screening visit or previous participation in this study.
* Participation in any nutritional study within 6 months prior to the screening visit.
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder
* Health conditions affecting food metabolism including food allergies, kidney disease, liver disease and/or gastrointestinal diseases.
* Use of concomitant medication that might interfere with the outcome of the study or increases the risk to the participant.
* Currently taking any other health food drinks/beverages or supplements (including nutritional supplements) or has been on supplements within a month prior to study start.
* Participant whose sibling is already a participant of this study.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Changes in regional brain hemodynamic response during attention, as measured by cognitive Functional Magnetic Resonance Imaging (fMRI) | From baseline to week 17
  Cognitive fMRI will be conducted at baseline and week 17 to assess the changes in regional brain hemodynamic response during attention task. Participants will be scanned while performing Sustained Attention to a Response Test (SART). During SART, a single digit (1-9) will be presented for 1 second(s). For first 333 miliseconds (ms), digit will be displayed in black font, then gray font for remaining 1s. Participants will be instructed to press a button when each digit turns gray. SART will have hard and easy block. During 'hard' block participants will be instructed to press the button for every digit except '3'. Whereas, during 'easy' block, they will be told that no 3's will be presented and no response needs to be withheld. Four easy blocks will be alternated with four hard blocks, with 15s rest between each. fMRI data will be acquired during the task and estimated by convolving hemodynamic response with task related brain Region of Interest

OTHER OUTCOMES:
Changes in regional brain hemodynamic response during working memory, as measured by cognitive fMRI | From baseline to week 17
  Cognitive fMRI will be conducted at baseline and week 17 to assess the changes regional brain hemodynamic response during working memory. The Participants will be scanned while performing n-back working memory task. They will be presented single digit number (0-9) one-by-one on the screen and will respond to targets and non-targets. Targets will be numbers that match those that occurred on the previous trial (1-back condition), the one before that (2-back condition) or the trial before that (3-back). A control condition will be responding to the target number ('0'). Each condition will be repeated thrice and the total task length will be about eight minutes. fMRI data will be acquired during the task and estimated by convolving hemodynamic response with task related brain ROI
Changes in functional hemodynamic response in cognitive network, as measured by resting-state fMRI | From baseline to week 17
  Resting state fMRI will be conducted at baseline and week 17 to determine functional connectivity between brain ROIs during resting state
Changes in gray matter density, as measured by structural MRI | From baseline to week 17
  Structural MRI will be conducted to define gray and white matter volumes. Changes in gray matter density will be measured at baseline and week 17
Correlation between performance scores on the Cambridge Neuropsychological Test Automated Battery (CANTAB) attention tasks and performance scores on the fMRI attention tasks | From baseline to week 17
  Rapid visual information processing test from CANTAB will be performed to assess sustained attention at baseline and week 17. The screen will display a box which randomly flashes the numbers 2-9. The participants will press the button on the screen when they see a target sequence of 3-5-7. The test will take approximately 7 min. Mean response data will be extracted and partial correlations accounting for agreed covariates will relate task performance on the CANTAB to the corresponding fMRI task response to assess brain-behavioral relationships
Correlation between performance scores on the CANTAB working memory tasks and performance scores on the fMRI working memory tasks | From baseline to week 17
  Spatial working memory test from CANTAB will be performed to assess working memory at baseline and week 17. The participants will search through a series of boxes until they find a blue chip. They will then move this blue chip to the "home" area on the right hand side of the screen. They will be told to look for the next blue chip which will not be in the same box as before. The number of boxes will be gradually increased from three to eight. Mean response data will be extracted and partial correlations accounting for agreed covariates will relate task performance on the CANTAB to the corresponding fMRI task response to assess brain-behavioral relationships
Correlation between the changes in regional brain hemodynamic response during working memory tasks, as measured using cognitive fMRI with the scores of working memory, as measured by the CANTAB | From baseline to week 17
  Partial correlations accounting for agreed covariates will be made to relate fMRI response on working memory task to the corresponding task performance on the CANTAB to assess brain-behavioral relationships at baseline and week 17
Correlation between changes in the regional brain hemodynamic response during attention tasks as measured using cognitive fMRI with the scores of attention, as measured by the CANTAB | From baseline to week 17
  Partial correlations accounting for agreed covariates will be made to relate fMRI response on working memory task to the corresponding task performance on the CANTAB to assess brain-behavioral relationships at baseline and week 17.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, New Delhi, India